CLINICAL TRIAL: NCT06152016
Title: BE FAST vs. FAST: A Randomized Trial Comparing Retention of Stroke Symptoms Between Two Mnemonics in the General Public.
Brief Title: BE FAST vs. FAST: A Study in the General Public.
Acronym: BFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: BayCare Health System (Other); Aurora BayCare Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 19-807
Record Dates: First submitted 2023-11-13; First posted 2023-11-30 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: BE-FAST; FAST
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BE-FAST (Other)
  Interventions: Other: BE-FAST
- FAST (Other)
  Interventions: Other: FAST

INTERVENTIONS:
Other: BE-FAST — This intervention includes those randomized to the education with the BE-FAST mnemonic.
  Arms: BE-FAST
Other: FAST — This intervention includes those randomized to the education with the FAST mnemonic.
  Arms: FAST

SUMMARY:
A randomized, blinded prospective study assessing retention of two stroke mnemonics (BE FAST and FAST) in the general public after receiving brief stroke education. Participants were randomized to one of two education arms and retention was tested at 3 different time intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Subject 18 years of age or older
2. Subject speaks English (Does not need interpreter)
3. Subject able to read English
4. Subject willing to provide a phone number for future follow up
5. Subject willing and agreeable to up to 2 phone follow up calls
6. Subject willing to provide verbal consent to participate

Exclusion Criteria:

1. Subject non-English speaking (needs interpreter)
2. Subject has visual or hearing impairment
3. Subject has history of Dementia or a learning disability
4. Subject had stroke education within the past year
5. Subject had a previous stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Recall Visit 1 | 60 minutes
  Number/percentage of participants in the FAST and BE-FAST groups at Visit 1 who accurately recall the mnemonic they were taught during the education session.

SECONDARY OUTCOMES:
Retention Rate Symptom | 30 days
  Retention rate of each stroke symptom in the mnemonic
Recall Rate Symptom | 30 days
  Total number of stroke symptoms that were accurately recalled by the participants
Recall Participant Percentage | 30 days
  Number/percentage of participants able to recall all the symptoms included in the mnemonic
Patrial Recall Participant Percentage | 30 days
  Number/percentage of participants able to recall 2 or more symptoms of the FAST mnemonic or 3 or more of the BE-FAST mnemonic.
Common Recall Participant Percentage | 30 days
  Number/percentage of participants able to recall the more common symptoms of each mnemonic (Facial weakness, arm weakness and speech difficulties)
Retention per Professional Background | 30 days
  Compare participants with medical vs. non-medical professional backgrounds and explore whether there are any group differences in retention rates.

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Darkhabani, MD, Principal Investigator — Aurora Baycare
Locations (1):
- Aurora BayCare Medical Center, Green Bay, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Darkhabani MZ, Homa-Bonell JK, Thoreson L, Bobholz JA, Spaulding D, Engebose M. BE FAST Versus FAST: A Randomized Pilot Trial Comparing Retention of Stroke Symptoms Between 2 Mnemonics. J Am Heart Assoc. 2024 Oct;13(19):e035696. doi: 10.1161/JAHA.123.035696. Epub 2024 Sep 18. PMID 39291473